CLINICAL TRIAL: NCT04704232
Title: Prospective,Double-blind,Randomized,Placebo-controlled Study of Safety,Efficacy, and Pharmacokinetics of Topical ACD440 in Healthy Volunteers
Brief Title: Study of Safety, Efficacy, and Pharmacokinetics of Topical ACD440 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AlzeCure Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D8000CI-001
Record Dates: First submitted 2020-12-22; First posted 2021-01-11 (Actual); Last update posted 2021-11-16 (Actual); Status verified 2021-11

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — 5'-palmitoyl cytarabine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACD440 (Active Comparator): Subjects are simultaneously exposed to topical administration of ACD440 in a crossover design in separate locations from the placebo exposure.
  Interventions: Drug: ACD440
- Placebo (Placebo Comparator): Subjects are simultaneously exposed to topical administration of placebo in a crossover design in separate locations from the ACD440 exposure.
  Interventions: Drug: PLAC

INTERVENTIONS:
Drug: ACD440 — Double blind, parallel within subject comparison
  Arms: ACD440
Drug: PLAC — Double blind, parallel within subject comparison
  Arms: Placebo

SUMMARY:
Phase 1 b placebo-controlled study in healthy volunteers to study safety, efficacy and pharmacokinetics of Topical ACD440 on normal skin, skin optimized for penetration and skin exposed to ultraviolet radiation

DETAILED DESCRIPTION:
This is an exploratory study, no primary or secondary endpoints are being defined.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteer
* Fitzpatrick skin type II or III
* Women not childbearing potential or highly effective contraception

Exclusion Criteria:

* Pregnancy, lactation
* Drug abuse
* Clinically significant illness
* Positive COVID 19 test at screening or COVID 19 infection in the past

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2021-01-12 (Actual); Primary Completion 2021-03-10 (Actual); Study Completion 2021-03-10 (Actual)

PRIMARY OUTCOMES:
Laser-evoked potentials as a tool for assessing the efficacy of antinociceptive drugs | 5 Days
  Not defined as primary as per protocol, but system does not seem to allow omittance of primaries

OTHER OUTCOMES:
Laser-evoked potentials as a tool for assessing the efficacy of antinociceptive drugs | 5 days
  Exploratory efficacy endpoint
Visual analog scale rating of laser induced pain | 5 days
  Exploratory efficacy endpoint
Number and percentage of subjects with adverse events | 5 days
  Safety endpoint
Number and percentage of subjects with clinically significant changes in 12-lead ECGs, vital signs and laboratory findings | 5 days
  Safety endpoint

CONTACTS AND LOCATIONS:
Locations (1):
- AlzeCure Pharma investigational site, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No